CLINICAL TRIAL: NCT04271787
Title: Periodontal Diseases Classification: Old is Gold or New is Bold
Brief Title: New Periodontal Classification
Status: Completed | Type: Observational
Sponsor: Beni-Suef University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Maha Abdelkawy, Phd, principle investigator, Beni-Suef University
Other Study IDs: FDBSUREC/27022019/AM
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Periodontal Diseases; Peri-Implantitis; Gingival Diseases
Keywords: Classification; Periodontal diseases; Periodontitis; Peri-implantitis
MeSH Terms: conditions — Periodontal Diseases; Peri-Implantitis; Gingival Diseases; Periodontitis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- strongly dissatisfied
  Interventions: Other: questionnaire
- dissatisfied
  Interventions: Other: questionnaire
- neutral
  Interventions: Other: questionnaire
- satisfied
  Interventions: Other: questionnaire
- strongly satisfied
  Interventions: Other: questionnaire
- don't know
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — Questionnaire

SUMMARY:
A new classification system of periodontal and peri-implant diseases and conditions was proposed by consensus of world experts in 2017. Since then there has been ongoing debates among periodontists regarding the application of the new classification. This study aims to shed light on the current understanding of the new classification among Egyptian periodontists.

DETAILED DESCRIPTION:
This study was approved by the Research Ethics Committee of Faculty of Dentistry Beni-Suef University (ID #FDBSUREC/27022019/AM) and was conducted in full accordance with the World Medical Association Declaration of Helsinki 1975, revised in 2003. The questionnaire was anonymous with no personal identification data. Completion and submission of the questionnaire was considered an approved informed consent to participate in the study by the Research Ethic Committee.

The questionnaire was designed by the authors and pilot tested among a group of 12 periodontists for validation. Afterwards, adjustments were made to ensure a clear and comprehensive version of the questionnaire. The questionnaire had a cover letter explaining the nature and purpose of the survey and comprised 15 questions. The first six statements of the questionnaire were descriptive in nature addressing the participant's demographics, and the seventh was a question whether the participant is aware of the new PDL classification or not. Only those who were aware of it were asked to proceed to 13 multiple choice questions using Likert scale; ranging from strongly disagree to strongly agree or from excellent to poor, in addition to "I don't know" option (8). There were also three open ended questions for further comments at the end of the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* periodontists

Exclusion Criteria:

* non periodontists

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: periodontists in various universities
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-11-04 (Actual)

PRIMARY OUTCOMES:
significant predictors of satisfaction with the new classification. | 4 months
  Binary logistic Regression analysis to determine significant predictors of new classification application. Ordinal Regression analysis to determine significant predictors of satisfaction with the new classification.

CONTACTS AND LOCATIONS:
Locations (1):
- Maha Abdelkawy, Phd, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
ONCE PUBLISHED
Supporting Information: SAP, ICF, CSR, Analytic Code
Time Frame: ONCE PUBLISHED